CLINICAL TRIAL: NCT00473655
Title: A Double-blind, Double Dummy, Phase IV, Randomized, Multicenter, Parallel Group, Placebo Controlled Trial to Evaluate the Effect of Rosuvastatin on Triglycerides Levels in Mexican Hypertriglyceridemic Patients
Brief Title: Effect of Rosuvastatin on Triglyceride Levels in Mexican Hypertriglyceridemic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DM-CRESTOR-0002
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Results first posted 2010-06-08 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-11

CONDITIONS: Hypertriglyceridemia; Hyperlipoproteinemia Type IV; Hyperlipoproteinemia Type V; Hyperlipoproteinemia Type IIb; Hyperlipidemia
Keywords: Triglycerides; hypertriglyceridemia; statins; rosuvastatin; hyperlipoproteinemia; Fredrickson Type IIb or IV
MeSH Terms: conditions — Hypertriglyceridemia; Hyperlipoproteinemia Type IV; Hyperlipoproteinemia Type V; Hyperlipoproteinemia Type II; Hyperlipidemias; Hyperlipoproteinemias | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: rosuvastatin — 10mg or 20mg

SUMMARY:
The primary purpose of this trial is to determine if the treatment with rosuvastatin 10 and 20mg/day during 8 weeks in hypertriglyceridemic patients will reduce their triglyceride levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years, both genders, without any previous treatment with statins or other lipid lowering drugs for at least 6 months
* With elevated triglycerides above 200 and below 800mg/dl and willing to follow all study procedures including assisting to clinics, fasting before blood samples and signing a written consent

Exclusion Criteria:

* High levels of low-density lipoprotein cholesterol (LDL-C)
* Unstable cardiovascular condition or awaiting a myocardial revascularization
* Congestive cardiac failure
* Uncontrolled diabetes
* Cancer
* Uncontrolled hypothyroidism
* Familial hypercholesterolemia
* Liver/muscle disease
* Pregnancy
* Other

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2007-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Polanco, MD, Study Director — AstraZeneca Mexico; Ana Polanco, MD, Study Chair — AstraZeneca Mexico; Juan Talavera, MD, Principal Investigator — IMSS
Locations (3):
- Mexico (3):
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo León

REFERENCES:
- [Derived] Talavera JO, Martinez G, Cervantes JL, Marin JA, Rodriguez-Briones I, Gonzalez JG, Ocampo R, Sanchez-Mijangos H, Bernal-Rosales LP, Polanco A. A double-blind, double-dummy, randomized, placebo-controlled trial to evaluate the effect of statin therapy on triglyceride levels in Mexican hypertriglyceridemic patients. Curr Med Res Opin. 2013 Apr;29(4):379-86. doi: 10.1185/03007995.2013.766590. Epub 2013 Feb 21. PMID 23323877

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants where outpatients recruited from clinical centers. Recruitment began on August 2007 and ends on October 2008
Pre-assignment Details: Participants with informed consent signed, and all inclusion criteria with no exclusion criteria, entered the lead in period, where they received a low fat diet. After 4 weeks if they still had TGs above 200 mg/dl they entered the randomization phase.
Groups:
- Rosuvastatin 10 mg: Rosuvastatin 10 mg
- Rosuvastatin 20 mg: Rosuvastatin 20 mg
- Placebo: Placebo
Period: Overall Study
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 20 mg | Placebo
Started | 111 (Just participants with TG above 200 mg/dl entered this period) | 112 (Just participants with TG above 200 mg/dl entered this period) | 111 (Just participants with TG above 200 mg/dl entered this period)
Completed | 102 (9 participants were lost of follow up) | 107 (5 participants were lost of follow up) | 103 (8 participants were lost of follow up)
Not Completed | 9 | 5 | 8
Not completed — Lost to Follow-up | 9 | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 20 mg | Placebo | Total
Number analyzed (Participants) | 111 | 112 | 111 | 334
Age Continuous [Mean (Standard Deviation); unit: Years]
  Age | 52.57 (12.77) | 53.14 (12) | 51.48 (13.47) | 52.4 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 67 | 54 | 173
  Male | 59 | 45 | 57 | 161
Arterial Hypertension [Number; unit: Participants]
  Arterial Hypertension | 36 | 35 | 34 | 105
Diabetes mellitus [Number; unit: Participants]
  Diabetes mellitus | 12 | 16 | 13 | 41
Body mass index continuous [Mean (Standard Deviation); unit: Kg/m2]
  Body mass index | 30.72 (5.11) | 29.77 (4.04) | 30.36 (4.90) | 30.28 (4.71)
HDL-C levels, continuous [Mean (Standard Deviation); unit: mg/dL]
  HDL-C | 33.50 (7.52) | 34.05 (6.88) | 32.30 (6.49) | 33.28 (6.99)
LDL-C, continuous [Mean (Standard Deviation); unit: mg/dL]
  LDL-C | 129.24 (28.23) | 130.51 (29.19) | 129.77 (31.10) | 129.84 (29.45)
TG levels, continuous [Mean (Standard Deviation); unit: mg/dL]
  Tg levels | 319.51 (131.95) | 296.78 (95.19) | 309.46 (99.55) | 308.25 (110.22)

OUTCOME MEASURES:

1. Primary Outcome: Change (Reduction) in Triglycerides Levels From Baseline to End of Treatment (Week 8)
Description: Reduction from baseline to end of study
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 101 | 107 | 103
mg/dL | 67.95 (128.46) | 78.61 (121.51) | 22.31 (120.54)

2. Secondary Outcome: Non-HDL-C Reduction
Description: Reduction from baseline to end of study
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 101 | 106 | 102
mg/dL | 52.76 (48.08) | 61.31 (46.63) | 1.06 (37.41)

3. Secondary Outcome: LDL-C Reduction
Description: Reduction from baseline to end of study
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 102 | 107 | 102
mg/dL | 42.23 (28.58) | 53.22 (32.80) | -2.66 (28.78)

4. Secondary Outcome: Total Cholesterol Reduction
Description: Reduction from baseline to end of study
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 102 | 107 | 103
mg/dL | 49.73 (41.13) | 63.32 (42.97) | -1.44 (34.98)

5. Secondary Outcome: HDL-C Increase
Description: Increase from baseline to end of study
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 101 | 104 | 102
mg/dL | 3.49 (7.16) | 2.49 (5.78) | 1.95 (7.42)

6. Secondary Outcome: ApoA1 Levels
Description: Change in the levels from baseline to end of study
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 101 | 106 | 102
mg/dl | 4.66 (23.38) | 6.79 (18.60) | 2.65 (19.40)

7. Secondary Outcome: hsCRP Reduction
Description: Reduction from baseline to end of study
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 102 | 107 | 103
mg/L | 0.19 (1.16) | 0.11 (0.35) | -0.01 (1.00)

8. Secondary Outcome: Adverse Events Reported
Description: Number of participants with AEs and SAEs reported
Time Frame: 8 weeks
Measure: Number; unit: Participants
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 111 | 112 | 111
Participants | 27 | 29 | 20

9. Secondary Outcome: ApoB Levels
Description: Change in the levels from baseline to end of study
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 20 mg | Placebo
Number analyzed (Participants) | 101 | 106 | 102
mg/dl | -27.05 (26.92) | -36.81 (23.51) | 1.43 (26.03)

ADVERSE EVENTS:
Arm/Group | Rosuvastatin 10 mg | Rosuvastatin 20 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/111 | 0/112 | 0/111
Other Adverse Events (participants affected / at risk) | 9/111 | 12/112 | 12/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 10 mg (N=111) | Rosuvastatin 20 mg (N=112) | Placebo (N=111)
Femur And Rotula Right Fracture That Required Hospitalization (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 10 mg (N=111) | Rosuvastatin 20 mg (N=112) | Placebo (N=111)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 5
Urinary tract infection (Renal and urinary disorders) | 1 | 1 | 3
Cephalea (Nervous system disorders) | 1 | 3 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pharyngotonsillitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Leg Edema (Renal and urinary disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI has the right to publish Study results in scientific journals. PI may use the Study results but not publish any results until: the date of the first Study results publication or the end of the 18-month period following the completion of the Study. PI shall provide AZ with the material for review. AZ has the right to publish the Study results